CLINICAL TRIAL: NCT03808233
Title: Reliability and Validity of the ACTIVE-mini for Quantifying Movement in Infants With Spinal Muscular Atrophy
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STU 052016-109
Record Dates: First submitted 2018-06-29; First posted 2019-01-17 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spinal Muscular Atrophy Type 1: Non rolling infants or children with SMA
  Interventions: Other: ACTIVE mini
- Non Rolling Function matched control: Non rolling typically developing infant
  Interventions: Other: ACTIVE mini

INTERVENTIONS:
Other: ACTIVE mini — the ACTIVE-mini, is a non-invasive method of recording movement in an infant using a KINECT camera system. This camera is positioned over a resting infant and measures natural movement over a two minute time period.

SUMMARY:
The purpose of this study is to investigate the measurement properties of the Ability Captured Through Interactive Video Evaluation-mini (ACTIVE-mini) for quantifying movement in infants with Spinal Muscular Atrophy (SMA). Specifically, I will investigate within-day and between-day test-retest reliability and calculate the minimal detectable change of the ACTIVE-mini. Additionally, I will determine the concurrent validity of the ACTIVE-mini with The Children's Hospital of Philadelphia Infant Test for Neuromuscular Disease (CHOP INTEND) and the construct validity of the ACTIVE-mini in infants with SMA using a known group methodology.

DETAILED DESCRIPTION:
This study was a cross-sectional, repeated measure design, investigating the test-retest within- and between-day reliability and the convergent construct validity and the known-groups method construct validity of the ACTIVE-mini. The group variable included two levels (non-rolling infants with SMA and function matched non-rolling typically developing infants). The dependent variables included a predicted CHOP INTEND score determined by data captured by the ACTIVE-mini and the CHOP INTEND extremity score. The dependent variables were collected at two time points over two days at a minimum of 24 hours and no more than 30 days between collections. Variables were collected in a standard order of assessment. All participants underwent all assessments as set out in the procedures. Based on results from pilot data, the conclusion was made that the ACTIVE-mini could quantify infant movement parameters well enough to warrant further investigation. These data were important in establishing the feasibility of the specific aims of this research, because they provide initial validation of the ability of ACTIVE-mini to quantify basic infant movement parameters

ELIGIBILITY:
Inclusion Criteria:

-

Participants will be included in this study if they:

* are non-rolling at time of enrollment
* age birth to 25 months
* have no concomitant system pathology that would limit clinical evaluation.

These inclusion criteria are set for both affected babies and healthy controls.

Exclusion Criteria:

Participants will be excluded from this study if they:

* demonstrate evidence of renal dysfunction, central nervous system damage, neuro-degenerative or neuromuscular disease other than SMA type I or II;
* require mechanical ventilation of any type > 16 hours per day.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: SMA
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-11-05 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
ACTIVE mini | 2 minutes
  the ACTIVE-mini, is a physiological parameter non-invasive method of recording movement in an infant using a KINECT camera system. This camera is positioned over a resting infant and measures natural movement over a two minute time period.

IPD SHARING:
Plan to Share IPD: No